CLINICAL TRIAL: NCT05000060
Title: A Prospective Randomized Open-Label Blinded Endpoint (PROBE) Pilot Trial of Early Restarting Antiplatelet Therapy Versus Usual Care After Traumatic Intracranial Hemorrhage.
Brief Title: Restart TICrH AP Pilot Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Truman J Milling Jr, Research Director SDMS Stroke Institute, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UT 101
Record Dates: First submitted 2021-07-26; First posted 2021-08-11 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Traumatic Intracranial Hemorrhage
Keywords: restart; antiplatelet; traumatic intracranial hemorrhage
MeSH Terms: conditions — Intracranial Hemorrhage, Traumatic

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Open Label Blinded Endpoint pilot trial of 100 patients
Who Masked: Outcomes Assessor
Masking Description: Blinded assessment and adjudication of endpoints
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 week restart (Experimental): Restart of mono or dual antiplatelet therapy one week post injury in TICrH patients
  Interventions: Other: Timing/1 week
- 3 week restart (Active Comparator): Usual Care for restart of mono or dual antiplatelet therapy after TICrH at clinician's discretion
  Interventions: Other: Timing/3 weeks

INTERVENTIONS:
Other: Timing/1 week — Time of restart of antiplatelet therapy is one week after injury
  Arms: 1 week restart
Other: Timing/3 weeks — Time of restart of antiplatelet therapy is left to treating clinician discretion
  Arms: 3 week restart

SUMMARY:
A Prospective Randomized Open-Label Blinded Endpoint (PROBE) Pilot Trial of restarting antiplatelet therapy at 1 week versus 3 weeks after traumatic intracranial hemorrhage with a primary composite endpoint of major bleeding and vascular occlusive events.

ELIGIBILITY:
Inclusion Criteria:

1. Acute traumatic intracranial hemorrhage on either mono or dual antiplatelet therapy
2. History of stroke, vascular stent or coronary or peripheral arterial disease as indication for antiplatelet *Restarting dual platelet therapy requires one of the following indications: 1) Acute myocardial infarction in the last year; 2) Coronary stent in the last year; 3) Non-cardioembolic stroke in the last 21 days (with switch to monotherapy at 21 days post stroke) 4) Peripheral arterial stent in the past month (with switch to monotherapy at one month post stent placement).

Exclusion Criteria:

1. SDH >8 mm maximum width or any midline shift at any time point or more than one SDH
2. Physician plan to start/restart anticoagulant therapy during trial period
3. Abbreviated Injury Scale other than head >3
4. Pregnancy
5. Inability to understand need for adherence to study protocol
6. Any active pathological bleeding (no acute blood on most recent CT)
7. Hypersensitivity to drug or other label contraindication
8. Any bleeding that the investigator deems unsafe to restart at 1 week post injury
9. Inability to swallow

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
major bleeding | 60 days
  Recurrent ICrH or other major bleeding defined by BARC3A
Major Vascular Occlusive events | Baseline (gambles performed pre-randomization)
  Ischemic stroke; myocardial infarction; mesenteric ischemia; peripheral arterial occlusion; deep vein thrombosis; pulmonary embolism; and carotid, coronary, or peripheral arterial revascularization procedures. Major vascular events defined by the Antithrombotic Trialists' Collaboration

IPD SHARING:
Plan to Share IPD: Yes
Data sharing with NIH BIOLINCC
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 years from study launch
Access Criteria: per NIH policy
URL: https://biolincc.nhlbi.nih.gov/home/